CLINICAL TRIAL: NCT05782153
Title: Comparing Self-Fitting Strategies in the Lexie Powered by Bose Hearing Aids: A Randomized Control Trial
Brief Title: Comparing Self-Fitting Strategies in the Lexie Powered by Bose Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: hearX Group (Industry)
Responsible Party: Principal Investigator, De Wet Swanepoel, Scientific advisor, hearX Group
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LexieB2PoweredbyBose
Record Dates: First submitted 2023-02-23; First posted 2023-03-23 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hearing Loss
Keywords: hearing loss; hearing aid; hearing rehabilitation; self-fitting hearing aid
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Cross-over within-subjects design. Forty participants will randomly be assigned to do a hearing aid self-fitting with direct adjustment (Intervention A) or a hearing aid self-fitting with in-situ audiometry (Intervention B) using the Lexie Powered by Bose hearing aids and will be asked to wear the hearing aids for four weeks. After four weeks, they will be crossed over to be fitted with the alternative fitting strategy, and they will be asked to wear the hearing aids again for four weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention A (hearing aid self-fitting with direct adjustment) (Active Comparator)
  Interventions: Device: Intervention A (hearing aid self-fitting with direct adjustment)
- Intervention B (hearing aid self-fitting with in-situ fitting) (Active Comparator)
  Interventions: Device: Intervention B (hearing aid self-fitting with in-situ fitting)

INTERVENTIONS:
Device: Intervention A (hearing aid self-fitting with direct adjustment) — The intervention offered is a hearing aid fitting with the Lexie B2 Powered by Bose receiver-in-the-canal hearing aids using a self-fitting strategy with direct adjustment. The hearing aids will be accompanied and operated with the Lexie smartphone application. Participants will complete a hearing screening (at 500, 1000, 2000 and 4000 Hz) called Hearing Check on the Lexie smartphone application, which will be used to tune the hearing aids according to frequency and loudness level. Participants will be able to use two wheels to change the loudness and fine-tune the hearing aids. Participants will wear the hearing aids for four weeks.
  Arms: Intervention A (hearing aid self-fitting with direct adjustment)
Device: Intervention B (hearing aid self-fitting with in-situ fitting) — The intervention offered is a hearing aid fitting with the Lexie B2 Powered by Bose receiver-in-the-canal hearing aids using the in-situ audiometry fitting strategy. The hearing aids will be accompanied and operated with the Lexie smartphone application. Participants will complete an in-situ audiogram on the Lexie app, which enables the measurement of hearing thresholds through the hearing aids (at 500, 1000, 2000 and 4000 Hz). The hearing aids will then be self-programmed according to the participant's in-situ audiogram with a proprietary fitting algorithm that is based on NAL-NL2. Participants will wear the hearing aids for four weeks.
  Arms: Intervention B (hearing aid self-fitting with in-situ fitting)

SUMMARY:
More than 1.5 billion people around the world experience hearing loss, of whom at least 430 million experience disabling hearing loss that will require rehabilitation. The majority of people have mild to moderate hearing loss and can benefit from hearing aids. However, hearing aid adoption around the world has been low, with global hearing aid coverage being less than 11%. This is partly due to limited access to hearing healthcare services and the high cost of hearing devices.

However, there have been significant efforts to improve access to hearing healthcare services. This includes rapid advances in hearing aids and new service-delivery models leading to more affordable and accessible options such as Over-the-Counter (OTC) hearing aids. On the 17th of October 2022, the Food and Drug Administration (FDA) established a regulatory category for OTC hearing aids. The final rule allows consumers with perceived mild to moderate hearing impairment to purchase hearing aids directly from stores or online retailers without the need for a medical exam, prescription or a fitting by an audiologist. The FDA defined two sub-categories for OTC hearing aids, namely 1) OTC hearing aids with standardized output profiles (i.e., pre-set programs) and 2) self-fitting OTC hearing aids which allow users to program their hearing aids with a self-fitting strategy and also customize their hearing aid settings according to their needs and preferences.

Sabin et al. (2020) was the first study to validate a self-fitting method using the Bose prototype hearing aid. This self-fitting method allowed users to select their own signal processing parameters using a mobile application consisting of two wheels that simultaneously control the gain and compression of all frequency bands. Sabin et al. (2020) evaluated the real-world performance of this approach by comparing gain, sound quality and clinical measures of hearing aid benefit and satisfaction between a group using the self-fitting method and a group that was professionally fitted with the same hearing aid. The gain selected by the self-fit group was within 1.8 dB overall and 5.6 dB per band compared to the gain selected by the audiologist. Participants in the self-fit group reported better sound quality, and there were no differences in clinical measures of hearing aid benefit or satisfaction.

Although a number of studies have compared self-fitting OTC devices to conventional hearing aids fitted by hearing healthcare professionals, no study has compared different self-fitting strategies in the same OTC device. Therefore, this study aims to compare the existing self-fitting strategy of the Lexie Powered by Bose hearing aids (i.e., direct adjustment) to a recently validated in-situ audiometry fitting strategy. The in-situ audiometry fitting strategy consists of in-situ thresholds measurements conducted at 500, 1000, 2000 and 4000 Hz through the hearing aids, which will be used with a proprietary fitting algorithm that is based on National Acoustics Laboratories' Non-Linear Version 2 (NAL-NL2) to self-program the hearing aids.

DETAILED DESCRIPTION:
* Objective: To compare an in-situ audiometry self-fitting strategy to the Bose self-fitting strategy (i.e., direct adjustment) using the same Lexie B2 Powered by Bose hearing aids. Hearing aid benefit and satisfaction will be compared in the same participants between the two fitting strategies. Additionally, Real Ear Measurements (REM) and speech perception will be compared in the same participants between the two fitting strategies.
* Hypothesis: The investigators hypothesize that there will be no statistically significant difference in terms of perceived hearing aid benefit and satisfaction, REM and speech perception within the same individual after receiving intervention A (hearing aid self-fitting with direct adjustment) and intervention B (hearing aid self-fitting with in-situ fitting) in a randomized, double-blind, cross-over within-subjects controlled trial.
* Design: Randomized, double-blind, cross-over within-subject controlled trial comparing an in-situ audiometry self-fitting strategy to the Bose self-fitting strategy (i.e., direct adjustment) using the same Lexie B2 Powered by Bose hearing aids in the same participants, which allows for participants to be their own control (n=40).
* Setting: This study will involve clinical audiometric testing at the Department of Speech-Language Pathology and Audiology, University of Pretoria, as well as a user field trial of the fitted hearing aids using each fitting strategy.
* Participants: Eligible participants will include 40 adults (>18 years) with a self-perceived mild-to-moderate level of hearing loss, without symptoms of outer- and middle ear pathology and who own a smartphone with access to mobile data (Android or iOS). Participants will be recruited and will randomly be assigned to a group using computer-generated randomization by an independent research assistant after being stratified for sex and degree of hearing loss.
* Intervention: Forty participants will randomly be assigned to be fitted with intervention A (hearing aid self-fitting with direct adjustment) or intervention B (hearing aid self-fitting with in-situ fitting) and wear the hearing aids for four weeks. After four weeks, they will be crossed over to be fitted with the alternative fitting strategy, and they will wear the hearing aids again for four weeks.
* Outcome measures: The primary outcome measure will be the Abbreviated Profile of Hearing Aid Benefit (APHAB). The secondary outcome measures will be the International Outcome Inventory for Hearing Aids (IOI-HA), Overall experience rating, REM, the QuickSIN speech-in-noise test and the Digits-in-noise test.

ELIGIBILITY:
Inclusion criteria:

1. Adults (>18 years) living in South Africa
2. Good English proficiency (measured using an online English proficiency test as well as self-report of English speaking competence)
3. Must have mild-to-moderate self-perceived hearing difficulties
4. Possession of a smartphone compatible with the Lexie app (iOS or Android)
5. Access to mobile data to operate the Lexie app
6. Must have transport to visit the initial and follow-up assessments

Exclusion criteria:

1. Normal hearing or self-perceived severe-to-profound hearing loss
2. Active outer or middle ear pathology
3. Poor English proficiency
4. Diagnosed cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline Abbreviated Profile of Hearing Aid Benefit (APHAB) | Baseline; After 4 weeks of field use with the first intervention; after 4 weeks of field use with the second intervention
  APHAB is a 24-item self-assessment inventory in which patients report the amount of trouble they experience hearing and communicating in noise in different everyday listening environments. The benefit is calculated by comparing the patient's reported difficulty in the unaided condition with their amount of difficulty when using amplification. The APHAB produces scores for 4 subscales: Ease of Communication (EC), Reverberation (RV), Background Noise (BN), and Aversiveness (AV).

SECONDARY OUTCOMES:
International Outcome Inventory for Hearing Aids (IOI-HA) | After 4 weeks of field use with the first intervention; after 4 weeks of field use with the second intervention
  IOI HA is a seven-item questionnaire designed to evaluate the effectiveness of hearing aid treatment. The responses of the items are assigned a value of 1 to 5, with higher scores indicating a more favourable outcome.
Overall experience rating | After first fitting; after second fitting
  In this questionnaire, participants will be asked about their overall experience with the hearing aid fitting and to rate how easy the process was using a Likert scale.
Change from baseline QuickSIN speech in noise test | Baseline; After 4 weeks of field use with the first intervention; after 4 weeks of field use with the second intervention
  The QuickSIN measures a person's ability to accurately hear speech in noise by determining a signal-to-noise ratio loss. A list of six sentences with five keywords per sentence is presented in four-talker babble noise. The sentences are presented at pre-recorded signal-to-noise ratios which decrease in 5-dB steps from 25 (very easy) to 0 (extremely difficult). The SNRs used are 25, 20, 15, 10, 5 and 0, encompassing normal to severely impaired performance in noise.
Change from baseline Digits-in-noise test (DIN) | Baseline; After 4 weeks of field use with the first intervention; after 4 weeks of field use with the second intervention
  The DIN measure primarily the auditory, or bottom-up, speech recognition abilities in noise. The test determines a speech reception threshold by presenting spoken digit triplets (e.g., 3-4-7) in speech-weighted background masking noise. Twenty-three digits are presented adaptively at different signal-to-noise ratios, based on correct or incorrect recognition of the digits. The speech reception threshold is determined by averaging the signal-to-noise ratios of the last 19-digit triplets.
Change from baseline Real-ear Measurements (REMs) | Baseline; Before and after 4 weeks of field use with the first intervention; before and after 4 weeks of field use with the second intervention
  REM involves placing a fine probe microphone into the ear canal to measure the sound at the eardrum. The hearing aid will be inserted in the ear alongside the probe microphone to measure the amplification effect within the patient's ear, taking into account the patient's ear acoustics.

CONTACTS AND LOCATIONS:
Overall Officials: De Wet Swanepoel, Principal Investigator — Department of Speech-Language Pathology and Audiology, University of Pretoria
Locations (1):
- University of Pretoria, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bisgaard N, Zimmer S, Laureyns M, Groth J. A model for estimating hearing aid coverage world-wide using historical data on hearing aid sales. Int J Audiol. 2022 Oct;61(10):841-849. doi: 10.1080/14992027.2021.1962551. Epub 2021 Aug 24. PMID 34428121
- [Background] Committee on Accessible and Affordable Hearing Health Care for Adults; Board on Health Sciences Policy; Health and Medicine Division; National Academies of Sciences, Engineering, and Medicine; Blazer DG, Domnitz S, Liverman CT, editors. Hearing Health Care for Adults: Priorities for Improving Access and Affordability. Washington (DC): National Academies Press (US); 2016 Sep 6. Available from http://www.ncbi.nlm.nih.gov/books/NBK367633/ PMID 27280276
- [Background] De Sousa KC, Manchaiah V, Moore DR, Graham MA, Swanepoel W. Effectiveness of an Over-the-Counter Self-fitting Hearing Aid Compared With an Audiologist-Fitted Hearing Aid: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Jun 1;149(6):522-530. doi: 10.1001/jamaoto.2023.0376. PMID 37052929
- [Background] Ferguson MA, Kitterick PT, Chong LY, Edmondson-Jones M, Barker F, Hoare DJ. Hearing aids for mild to moderate hearing loss in adults. Cochrane Database Syst Rev. 2017 Sep 25;9(9):CD012023. doi: 10.1002/14651858.CD012023.pub2. PMID 28944461
- [Background] Food and Drug Administration. (2021). Medical Devices; Ear, Nose, and Throat Devices; Establishing Over-the-Counter Hearing Aids. https://www.govinfo.gov/content/pkg/FR-2021-10-20/pdf/2021-22473.pdf
- [Background] Humes LE, Rogers SE, Quigley TM, Main AK, Kinney DL, Herring C. The Effects of Service-Delivery Model and Purchase Price on Hearing-Aid Outcomes in Older Adults: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Am J Audiol. 2017 Mar 1;26(1):53-79. doi: 10.1044/2017_AJA-16-0111. PMID 28252160
- [Background] Keidser G, Convery E. Outcomes With a Self-Fitting Hearing Aid. Trends Hear. 2018 Jan-Dec;22:2331216518768958. doi: 10.1177/2331216518768958. PMID 29716438
- [Background] Manchaiah V, Taylor B, Dockens AL, Tran NR, Lane K, Castle M, Grover V. Applications of direct-to-consumer hearing devices for adults with hearing loss: a review. Clin Interv Aging. 2017 May 18;12:859-871. doi: 10.2147/CIA.S135390. eCollection 2017. PMID 28553093
- [Background] Sabin AT, Van Tasell DJ, Rabinowitz B, Dhar S. Validation of a Self-Fitting Method for Over-the-Counter Hearing Aids. Trends Hear. 2020 Jan-Dec;24:2331216519900589. doi: 10.1177/2331216519900589. PMID 32003285
- [Background] Swanepoel W, Oosthuizen I, Graham MA, Manchaiah V. Comparing Hearing Aid Outcomes in Adults Using Over-the-Counter and Hearing Care Professional Service Delivery Models. Am J Audiol. 2023 Jun;32(2):314-322. doi: 10.1044/2022_AJA-22-00130. Epub 2023 Mar 6. PMID 36876936
- [Background] World Health Organization. (2021). World report on hearing. Retrieved from https://www.who.int/publications/i/item/world-report-on-hearing
- [Derived] Knoetze M, Manchaiah V, De Sousa K, Moore DR, Swanepoel W. Comparing Self-Fitting Strategies for Over-the-Counter Hearing Aids: A Crossover Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Sep 1;150(9):784-791. doi: 10.1001/jamaoto.2024.2007. PMID 39052241